CLINICAL TRIAL: NCT05529667
Title: An Open Label, Single-Arm, Multi-center Phase Ib/II Study to Evaluate the Safety and Efficacy of INCB054828 in Combination With Paclitaxel as a Second Line Treatment in Recurrent/Advanced Gastric Cancer With FGFs/FGFRs Genetic Aberration.
Brief Title: Fibroblast Growth Factor (FGFs) / Fibroblast Growth Factor Receptor (FGFRs) Genetic as a Second-line Therapy for Recurrent / Progressive Gastric Cancer With INCB054828 and Paclitaxel a Study to Evaluate the Safety and Efficacy of Combination Therapy.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2018-0327
Record Dates: First submitted 2022-08-16; First posted 2022-09-07 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Fibroblast Growth Factors (FGFs)/Fibroblast Growth Factor Receptors (FGFRs) Genetic Aberration Gastric Cancer, INCB054828, Paclitaxel
MeSH Terms: interventions — pemigatinib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): 1. phase>
     * INCB054828 begins with oral administration of 13.5 mg once a day.
     * Paclitaxel is administered intravenously every week at 80mg / m2. (Days 1, 8 and 15) It is one cycle of 4 weeks and it is administered until the time of disease progression.
  2. phase>
     * INCB54828 is dosed at the dose specified in phase 1.
     * Paclitaxel is administered intravenously every week at 80mg / m2. (Days 1, 8 and 15) It is one cycle of 4 weeks and it is administered until the time of disease progression
  Interventions: Drug: INCB054828, Paclitaxel

INTERVENTIONS:
Drug: INCB054828, Paclitaxel — phase 1>
  - Approximately 3-12 patients will be enrolled. The dose escalation will be three patients registered for each cohort until the first dose-limiting toxicity appears during the four weeks of treatment and observation.
  phase 2> Phase 2 studies will be extended to a total of 30 patients with a two-phase recommended dose. Patients will be treated until the time of disease progression, intolerable toxicity, rejection of the patient, or withdrawal of consent.

SUMMARY:
This study was conducted as a second-line treatment of recurrent / progressive gastric cancer patients with FGFs / FGFRs genetic mutations in the Ib / II clinical trial. The maximum maximal tolerated dose (MTD) and 2-phase recommended dose in combination with INCB054828 and paclitaxel (recommended phase II dose, RP2D), and evaluate the safety and clinical efficacy of this combination therapy. This study consists of two steps: Phase 1 is a dose escalation study to determine the maximum tolerated dose and 2-phase recommended dose of weekly paclitaxel and INCB054828 combination therapy, and Phase 2 is the dose escalation study in combination with INCB054828 and paclitaxel Assess safety and tolerability and identify antitumor effects in stomach cancer with FGFs / FGFRs genetic mutations.

DETAILED DESCRIPTION:
1. phase>

   - Approximately 3-12 patients will be enrolled. The dose escalation will be three patients registered for each cohort until the first dose-limiting toxicity appears during the four weeks of treatment and observation. 13.5mg, once a day begins to take. The paclitaxel is administered once a week for three consecutive weeks and then for one week, followed by a total of four weeks in one cycle.
2. phase> Phase 2 studies will be extended to a total of 30 patients with a two-phase recommended dose. Patients will be treated until the time of disease progression, intolerable toxicity, rejection of the patient, or withdrawal of consent. In its pre-screening phase, its next generation sequencing (NGS) is performed. Patients with FGFs / FGFRs genetic abnormalities may be enrolled in this study. If a patient has multiple genetic abnormalities, he or she will first be enrolled in a treatment group that targets a rare genetic abnormality. Registered patients will be treated on a continuous basis every four weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who agreed in writing to the clinical study consent
2. Histologically or cytologically confirmed advanced gastric adenocarcinoma. Patients must have experienced objective radiological or disease progress with evidence during or after primary therapy with fluoropyrimidine and platinum.
3. FGFs / FGFRs have genetic variation on NGS.
4. Patients whose life expectancy is at least 3 months
5. If the Eastern Cooperative Oncology Group (ECOG) is 0 or 1
6. Measurable or assessable lesion based on RECIST 1.1 scale
7. Must be swallowed, should be able to take oral medication
8. Possible long-term function to receive chemotherapy.
9. Patients receiving anti-HER2 therapy for HER2 negative or HER2-positive primary treatment

Exclusion Criteria:

1. When chemotherapy exceeded the first treatment
2. Patients with multiple cancers
3. Severe hypersensitivity reactions to anti-FGFR2 agents either now or in the past
4. Patients with endocrine metabolic syndrome or history of calcium-phosphate homeostasis
5. Patients with ectopic neoplasm or history of soft tissue, kidney, large intestine, heart, or abdomen
6. Corneal lesions such as bullous keratopathy, corneal erosion, corneal erosion, corneal ulcer, corneal inflammation and keratoconjunctivitis were confirmed by ophthalmic examination
7. Patients with metastasis to the brain or meninges. However, patients who do not have symptoms and do not need treatment can register.
8. Clinically significant digestive system problems that can cause abnormalities in taking or absorbing clinical drugs
9. Patients with uncontrollable or significant cardiovascular disease
10. Patients with systemic infections requiring treatment
11. Patients who were exposed to paclitaxel at or before the taxane
12. If you undergo major surgery within 28 days before enrollment for this trial
13. Patients who received radiotherapy for gastric cancer within 28 days prior to enrollment for this trial. However, the investigation of bone turnover was conducted within 14 days before the registration for this trial
14. If you received general chemotherapy within 14 days of enrollment for this trial
15. Patients who are positive for human immunodeficiency virus (HIV-1) antibody test,
16. HBsAg results positive, HBV viral load greater than 2000 IU / ml (104 copies / ml), or HCV antibody test positive
17. Patients who are pregnant, lactating, or are likely to be pregnant
18. Anemia and hair loss are excluded if previous chemotherapy treatment has toxicity that is not recovered below grade 2.
19. Patients who are judged to have lost their ability to cope with dementia or other comorbid conditions
20. Other Patients who the examiner or the examiner deemed inappropriate for the clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
MTD | 4 weeks
  Part 1, Phase Ib Maximum Tolerated dose (MTD)
Recommended phase 2 dose (RP2D) | 4 weeks
  Part 1, Phase Ib Recommended phase 2 dose as determined by Dose limiting Toxicity (DLT).
PFS | 24 weeks
  Prart 2, Phase II Progression-free survival (PFS): PFS is defined as the interval between the date of first dose and the earliest date of disease progression or death due to any cause.

SECONDARY OUTCOMES:
ORR | 3 years
  Objective Response Rate (ORR): The duration of response. ORR is defined as the percentage of subjects with a confirmed CR or PR per RECIST v1.1
DCR | 3 years
  Disease Control Rate (DCR): DCR is the proportion of randomized patients achieving a best overall response of CR, PR, or SD.
OS | 3 years
  Overall Survival (OS): OS is the time from the date of first dose and the date of death from any cause.
Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | 3 years
  Safety and tolerability of the Varlitinib and Paclitaxel combination therapy as determined by: adverse events (categorized in accordance with CTCAE 4.03).

CONTACTS AND LOCATIONS:
Overall Officials: SUN YOUNG RHA, Principal Investigator — Yonsei Cancer Center, Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No